CLINICAL TRIAL: NCT00247091
Title: Impact of HIV on Measles and Measles Immunisation
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Burroughs Wellcome (Industry); London School of Hygiene and Tropical Medicine (Other); University of Zambia (Other)
Other Study IDs: GR059114MA
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2005-11-01 (Estimated); Status verified 2005-10

CONDITIONS: HIV Infection; Measles; Children
Keywords: HIV; measles; measles vaccine; children; Zambia
MeSH Terms: conditions — HIV Infections; Measles

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Biological: standard-titer measles vaccine

SUMMARY:
We conducted a longitudinal study to assess the immunogenicity of standard-titer measles vaccine in HIV-infected and uninfected Zambian children. The study hypothesis was that HIV-infected children would have higher rates of primary and secondary measles vaccine failure compared to uninfected children, contributing to decreased levels of population immunity to measles and facilitating measles virus transmission in regions of high HIV prevalence.

DETAILED DESCRIPTION:
Despite great progress in measles control in sub-Saharan Africa, measles remains a significant cause of morbidity and mortality in young children. In regions of high HIV prevalence, measles virus transmission may be sustained despite high immunization coverage rates if HIV-infected children are important transmitters of measles virus. Factors potentially contributing to enhanced measles virus transmission by HIV-infected children include an early decline in protective maternal antibody titers resulting in susceptibility to measles at a younger age, and high rates of primary and secondary measles vaccine failure. To evaluate the potential impact of the HIV-1 epidemic on immunity following measles vaccination, we conducted a longitudinal study to compare the primary vaccine failure rate and rate of antibody decline following administration of standard-titer measles vaccine at nine months of age to HIV-infected and HIV-uninfected Zambian children. Our results show that children born to HIV-infected women have lower levels of passively-acquired maternal antibodies to measles virus prior to the age of routine vaccination at 9 months, and HIV-infected children are particularly susceptible to measles in infancy. This finding supports the WHO recommendation to provide the first dose of measles vaccine to HIV-infected children at 6 months. Furthermore, HIV-infected children develop adequate primary antibody responses to measles vaccine in the months following vaccination but lose protective antibody titers by two to three years of age. Mitigating the potential impact of this decreased immunogenicity on the level of population immunity to measles virus was the high mortality rate observed among HIV-infected children. Improved access to antiretroviral therapy will likely improve the survival of HIV-infected children without enhancing protective immunity to measles virus, although this has yet to be investigated. We are working to incorporate our findings into a mathematical model to better understand the impact of the HIV-1 epidemic on measles control strategies and to investigate the immunologic mechanisms for impaired memory B cell responses in HIV-infected children.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2 to 8 months presenting for well-child care
* reside within 10 miles of the study clinic
* parents or caretakers provide signed informed consent

Exclusion Criteria:

-children with severe illness

Ages: 2 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700
Dates: Start 2000-05; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: William J. Moss, MD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; Felicity Cutts, MD, Principal Investigator — London School of Hygiene and Tropical Medicine; Francis Kasolo, MD, PhD, Principal Investigator — University of Zambia
Locations (1):
- Chawama Clinic, Lusaka, Zambia